CLINICAL TRIAL: NCT03048084
Title: Seizure Treatment in Glioma (STING): Comparing a Treatment Strategy with Levetiracetam Versus Treatment with Valproic Acid in Glioma Patients with a First Seizure
Brief Title: Seizure Treatment in Glioma
Acronym: STING
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Medical Center Haaglanden (Other); Erasmus Medical Center (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, j.a.f.koekkoek, MD PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 77353
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Levetiracetam; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levetiracetam (Active Comparator): Patients in this treatment arm will receive levetiracetam monotherapy. The dosage depends on the specific treatment step, as indicated in the protocol. In step 1, patients will receive 2x500 mg/d levetiracetam in the form of tablets. In step 2, dosage is increased to 1x250 plus 1x500 mg/d and in step 3 to 2x1000 mg/d levetiracetam. In step 4, levetiracetam is increased to 2x1500mg/d. In the fifth treatment step, patients will receive 2x1500 mg/d levetiracetam, and another AED will be added. The type and dosage of this add-on AED is according to the physician's preference, but in line with current clinical practice in the Netherlands.
  Interventions: Drug: Levetiracetam
- Valproic acid (Active Comparator): Patients in this treatment arm will receive valproic acid monotherapy. The dosage depends on the specific treatment step, as indicated in the protocol. In step 1, patients will receive 2x500 mg/d valproic acid in the form of tablets. In step 2, dosage is increased to 1x250 plus 1x500 mg/d and in step 3 to 2x1000 mg/d valproic acid. In step 4, valproic acid dosage is increased to a maximum of 2x1250mg/d. In the fifth treatment step, patients will receive 2x1250mg valproic acid, and another AED will be added. The type and dosage of this add-on AED is according to the physician's preference, but in line with current clinical practice in the Netherlands.
  Interventions: Drug: Valproic Acid

INTERVENTIONS:
Drug: Levetiracetam — Antiepileptic drug levetiracetam
  Other Names: Keppra
  Arms: Levetiracetam
Drug: Valproic Acid — Antiepileptic drug valproic acid
  Other Names: Depakine
  Arms: Valproic acid

SUMMARY:
Currently, treatment with a specific anti-epileptic drug mainly depends on the physicians' preference, as there are no studies supporting the use of one specific anticonvulsant in glioma patients. The overall aim of this randomized controlled trial is to directly compare the effectiveness of treatment with levetiracetam or valproic acid in glioma patients with a first seizure.

DETAILED DESCRIPTION:
Currently, treatment of glioma patients with a specific anti-epileptic drug (AED) mainly depends on the physicians' preference, as there is no robust evidence from randomized controlled trials supporting the use of one specific anticonvulsant above the other in glioma patients.

Levetiracetam and valproic acid are the most commonly used AEDs in glioma patients. Both drugs are used for the treatment of seizures, have similar toxicity profiles and are non-enzyme inducing AEDs, therefore not interfering with chemotherapeutic drugs. However, it is not known whether one drug is more effective than the other in reducing seizures.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven or suspected diffuse astrocytoma (Isocytrate Dehydrogenase-1 (IDH-1) wildtype or IDH-1 mutated), diffuse oligodendroglioma (IDH-1 mutated and 1p/19q co-deleted), anaplastic astrocytoma (IDH-1 wildtype or IDH-1 mutated), anaplastic oligodendroglioma (IDH-1 mutated and 1p/19q co-deleted), glioblastoma (IDH-1 wild-type or IDH-1 mutated), or diffuse astrocytoma not otherwise specified (NOS), anaplastic astrocytoma NOS, oligodendroglioma NOS, oligoastrocytoma NOS, anaplastic oligoastrocytoma NOS, anaplastic oligodendroglioma NOS or glioblastoma NOS.
* Adult patients: ≥18 years of age
* First epileptic seizure, no longer than 2 weeks ago
* Monotherapy with antiepileptic drugs is considered most appropriate at the time of randomization
* Willing to provide written informed consent

Exclusion Criteria:

* Previously treated with antiepileptic drugs, except emergency treatment in the past 2 weeks
* History of non-brain tumor related epilepsy
* Pregnancy
* Presence of contra-indications for use of levetiracetam or valproic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Ongoing seizure freedom at 6 months | 6 months
  The percentage of patients with ongoing seizure freedom at 6 months

SECONDARY OUTCOMES:
Time to 6 months seizure freedom | 0, 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months or 0, 1, 6, 12, 18, 24 and 30 months, depending on a 3-monthly or 6-monthly follow-up schedule respectively
  Time to 6 months seizure freedom
Seizure outcome at 12 months | 12 months
  Seizure outcome at 12 months
Adverse effects of the treatment | 0, 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months or 0, 1, 6, 12, 18, 24 and 30 months, depending on a 3-monthly or 6-monthly follow-up schedule respectively
  Adverse effects of the treatment
Hospitalisation rate | 0, 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months or 0, 1, 6, 12, 18, 24 and 30 months, depending on a 3-monthly or 6-monthly follow-up schedule respectively
  hospitalization rate due to treatment failure
Health-related quality of life | 0, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months or 0, 6, 12, 18, 24 and 30 months, depending on a 3-monthly or 6-monthly follow-up schedule respectively
  Health-related quality of life
Cognitive complaints | 0, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months or 0, 6, 12, 18, 24 and 30 months, depending on a 3-monthly or 6-monthly follow-up schedule respectively
  Cognitive complaints
Mood | 0, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months or 0, 6, 12, 18, 24 and 30 months, depending on a 3-monthly or 6-monthly follow-up schedule respectively
  Anxiety and depression
Performance Status | 0, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months or 0, 6, 12, 18, 24 and 30 months, depending on a 3-monthly or 6-monthly follow-up schedule respectively
  Karnofsky Performance Status Score
Epilepsy burden | 0, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months or 0, 6, 12, 18, 24 and 30 months, depending on a 3-monthly or 6-monthly follow-up schedule respectively
  Epilepsy burden
Treatment response | 0, 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months or 0, 1, 6, 12, 18, 24 and 30 months, depending on a 3-monthly or 6-monthly follow-up schedule respectively
  Treatment response (e.g., maximum dosage of AED, use of add-on AED)
Progression-free survival | 0, 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months or 0, 1, 6, 12, 18, 24 and 30 months, depending on a 3-monthly or 6-monthly follow-up schedule respectively
  Progression-free survival
Overall survival | 0, 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months or 0, 1, 6, 12, 18, 24 and 30 months, depending on a 3-monthly or 6-monthly follow-up schedule respectively
  Overall survival

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - Amsterdam UMC, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam
  - Haaglanden Medical Center, The Hague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Meer PB, Taphoorn MJB, Koekkoek JAF. Management of epilepsy in brain tumor patients. Curr Opin Oncol. 2022 Nov 1;34(6):685-690. doi: 10.1097/CCO.0000000000000876. Epub 2022 Jul 16. PMID 35838207
- [Derived] Lang F, Liu Y, Chou FJ, Yang C. Genotoxic therapy and resistance mechanism in gliomas. Pharmacol Ther. 2021 Dec;228:107922. doi: 10.1016/j.pharmthera.2021.107922. Epub 2021 Jun 23. PMID 34171339